CLINICAL TRIAL: NCT00643838
Title: Sedation Faisability by Inhalation of Kalinox 170 Bar During Therapeutic Cares in Primary Care Dental Centers
Brief Title: Use of 50% Nitrous Oxide / 50% Oxygen Premix in Primary Care Dental Centers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT : 2006-005691-40
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2009-01

CONDITIONS: Dental Cares

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Misture of 50% nitrous oxide and 50% oxygen
  Interventions: Drug: Kalinox 170 bar

INTERVENTIONS:
Drug: Kalinox 170 bar — Flow of gas administrated to the patient between 4 and 15 litre/min and less than 1 hour

SUMMARY:
A 50% nitrous oxide / 50% oxygen premix is administrated to the patient during the realization of dental cares. This openly clinical trial is done in 36 French primary care dental centers, especially on anxious and phobic patients but also on infants or mental deficient adults. At least 480 patients will be included in this clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* anxious and/or phobic patients having a vomiting reflex
* very young children requiring selective dental cares
* mental deficient patient
* patient having specific phobia linked to the dental care to be done
* patient from 1 year old
* ASA 1 or ASA 2 patient
* existing of efficient contraception

Exclusion Criteria:

* ASA 3 or ASA 4 patient
* patient already treated without using Kalinox's sedation
* patient already included in this protocol in a delay lower than 7 days
* contraindication linked to the experimental product
* Kalinox's inhalation duration higher than 1 hour
* pregnant or breast-feeding women

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Pain measurement by using Visual Analog Scale (VAS) and Face Pain Scale (FPS) | At the end of the dental care

SECONDARY OUTCOMES:
Patient's acceptance and doctor's satisfaction | At the end of dental care

CONTACTS AND LOCATIONS:
Locations (1):
- Primary dental care centers, Clermont-Ferrand, France

REFERENCES:
- [Result] Hennequin M, Collado V, Faulks D, Koscielny S, Onody P, Nicolas E. A clinical trial of efficacy and safety of inhalation sedation with a 50% nitrous oxide/oxygen premix (Kalinox) in general practice. Clin Oral Investig. 2012 Apr;16(2):633-42. doi: 10.1007/s00784-011-0550-y. Epub 2011 Mar 29. PMID 22186944